CLINICAL TRIAL: NCT07341620
Title: Effectiveness of an Online Interactive E-book in Enhancing Home Care Nurses' Knowledge, Perceived Barriers, and Self-efficacy in Home Pressure Injury Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Ching Lin, PhD student and Investigator, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KMUHIRB-F(I)-20250035
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pressure Injuries
Keywords: Home care nursing; home health nurses; pressure injuries; home health care; digital education
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive E-book on Pressure Injury Care (Experimental): Participants in this group will access an online interactive e-book focused on home-based pressure injury prevention and wound care for one month. The e-book consists of 11 interactive learning units.
  Interventions: Other: Interactive E-book on Pressure Injury Care
- MOHW Standard PDF Educational Materials (Active Comparator): Participants in this group will be provided with standard PDF educational materials on pressure injuries from the Ministry of Health and Welfare (MOHW) Long-term Care section for one month.
  Interventions: Other: MOHW Standard PDF Educational Materials

INTERVENTIONS:
Other: Interactive E-book on Pressure Injury Care — An online interactive digital e-book containing 11 units on pressure injury prevention and wound care management for home care nurses.
  Arms: Interactive E-book on Pressure Injury Care
Other: MOHW Standard PDF Educational Materials — Standardized PDF educational documents regarding pressure injuries provided by the Ministry of Health and Welfare (MOHW) Long-term Care section.
  Arms: MOHW Standard PDF Educational Materials

SUMMARY:
The goal of this study is to learn if an interactive e-book helps home care nurses improve their skills in managing pressure injuries at home. It will also learn if digital learning can overcome the challenges of traditional training. The main questions it aims to answer are:

1. Does the e-book increase home care nurses' knowledge about pressure injury prevention and treatment?
2. Does it improve their confidence and reduce the barriers they face when providing wound care?
3. How long do the learning benefits last after completing the program?

Researchers will compare an interactive e-book to standard PDF training materials from the Ministry of Health and Welfare (MOHW) to see which is more effective for nursing education.

Participants will:

1. Use an online interactive e-book covering 11 units of wound care for 1 month
2. Use standard PDF training materials from the MOHW Long-term Care section
3. Complete surveys about their knowledge and skills before the study, immediately after the program, and 1 month later

Expected Outcomes and Contributions:

This study aims to solve the problem of nursing shortages and training difficulties in rural areas. The researchers expect that home care nurses will become more competent in wound management, leading to better patient health and fewer hospital readmissions. These results will support Taiwan's "Long-term Care 3.0" policy by driving innovation in digital education.

DETAILED DESCRIPTION:
The goal of this study is to learn if an interactive e-book helps home care nurses improve their skills in managing pressure injuries at home. It will also learn if this digital tool can overcome barriers to traditional training.

The main questions it aims to answer are:

1. Does the e-book increase home care nurses' knowledge about pressure injury prevention and treatment?
2. Does it improve their confidence and reduce the barriers they face when providing wound care?
3. How long do these learning benefits last after the program ends? Researchers will compare an interactive e-book to standard PDF training materials from the Ministry of Health and Welfare (MOHW) to see which is more effective for nursing education.

Participants will:

1. Use an online interactive e-book on wound care for 1 month (Experimental Group)
2. Read standard PDF training materials from the MOHW Long-term Care section (Control Group)

Complete surveys about their knowledge and skills before the study, immediately after the program, and 1 month later

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses aged 18 years or older.
* Currently employed full-time as a home care nurse in a hospital-affiliated home care agency, private home care agency, or public health center.
* Have at least six months of clinical experience in home care nursing.
* Willing to participate in this study and sign the informed consent form.

Exclusion Criteria:

* Home care nurses who hold specialized certifications related to advanced wound care (due to their existing high level of expertise in pressure injury management).
* Nurses practicing in community nursing homes or residential care facilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Pressure Injury Knowledge Assessment Score (PUKAT 2.0) | Baseline (Pre-intervention), 1 month (immediately post-intervention), and 2 months (1-month follow-up).
  Evaluation of home care nurses' knowledge using the Pressure Ulcer Knowledge Assessment Tool (PUKAT 2.0). The tool assesses competency in prevention and management of pressure injuries.

SECONDARY OUTCOMES:
Perceived Barriers to Wound Care (WCBS) | Baseline (Pre-intervention), 1 month (immediately post-intervention), and 2 months (1-month follow-up).
  Measured by the Wound Care Perceived Barriers Scale (WCBS), consisting of 16 items. Each item is rated on a 5-point Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). Total scores range from 16 to 80 points. A higher score indicates that the participant perceives significantly greater barriers to performing wound care.
Pressure Ulcer Management Self-Efficacy (PUM-SES) | Baseline (Pre-intervention), 1 month (immediately post-intervention), and 2 months (1-month follow-up).
  Measured by the Pressure Ulcer Management Self-Efficacy Scale (PUM-SES). Each item is rated on a 5-point Likert scale from 1 (Totally Incapable) to 5 (Totally Capable). Total scores range from 10 to 50 points. A higher score indicates stronger self-efficacy in the prevention and management of pressure injuries.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant privacy and maintain data confidentiality as per the institutional review board requirements.